CLINICAL TRIAL: NCT06212440
Title: Clinical Application of Multi-modal Sentinel Lymph Node Staining Method in Breast Cancer Patients Who Receive Neoadjuvant Chemotherapy : Expanded Access Clinical Study in 3 Arms
Brief Title: Clinical Application of Multi-modal Sentinel Lymph Node Staining Method in Breast Cancer Patients After Neoadjuvant Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Seeyoun Lee, Doctor, M.D., head of center for breast cancer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010242-2
Record Dates: First submitted 2023-02-14; First posted 2024-01-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Sentinel Lymph Node Biopsy; Neoadjuvant Therapy; Breast Neoplasm
Keywords: breast cancer; sentinel node biopsy; neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: open-label, prospective, single-institution, 3-arms expended randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- RI + ICG-F (Experimental): Participants undergo sentinel lymph node biopsy using Radioactive Isotope (RI) and Indocyanine Green Fluorescence (ICG-F) for lymphatic mapping.
  Interventions: Diagnostic Test: Radioactive Isotope (RI) Mapping; Diagnostic Test: Indocyanine Green Fluorescence (ICG-F) Mapping
- RI + Vital Dye (Experimental): Participants undergo sentinel lymph node biopsy using Radioactive Isotope (RI) and Vital Dye for lymphatic mapping.
  Interventions: Diagnostic Test: Radioactive Isotope (RI) Mapping; Diagnostic Test: Vital Dye Mapping
- Vital Dye + ICG-F (Experimental): Participants undergo sentinel lymph node biopsy using Vital Dye and Indocyanine Green Fluorescence (ICG-F) for lymphatic mapping.
  Interventions: Diagnostic Test: Indocyanine Green Fluorescence (ICG-F) Mapping; Diagnostic Test: Vital Dye Mapping

INTERVENTIONS:
Diagnostic Test: Radioactive Isotope (RI) Mapping — Administered via peritumoral or subareolar injection for sentinel lymph node detection.
  Arms: RI + ICG-F; RI + Vital Dye
Diagnostic Test: Indocyanine Green Fluorescence (ICG-F) Mapping — Administered via peritumoral or subareolar injection, detected using near-infrared fluorescence imaging.
  Arms: RI + ICG-F; Vital Dye + ICG-F
Diagnostic Test: Vital Dye Mapping — Administered via peritumoral or subareolar injection for intraoperative visualization of lymphatic drainage pathways.
  Arms: RI + Vital Dye; Vital Dye + ICG-F

SUMMARY:
This clinical trial aimed to confirm the effectiveness of sentinel lymph node surgery by determining the lymph node identification rate using multimodal sentinel lymph node marker methods in patients with advanced breast cancer undergoing neoadjuvant chemotherapy (NAC).

DETAILED DESCRIPTION:
After NAC, the sentinel lymph node (SLN) identification rate is lower, and it has a higher false-negative rate than that in early-stage breast cancer. As appropriate SLN surgery directly affects the treatment and prognosis of patients undergoing NAC, evaluation to identify SLN using various methods is necessary.

This clinical trial aimed to confirm the effectiveness of sentinel lymph node surgery by determining the lymph node identification rate using multimodal sentinel lymph node marker methods in patients with advanced breast cancer undergoing neoadjuvant chemotherapy (NAC).

ELIGIBILITY:
Inclusion Criteria:

* The patient with locally advanced breast cancer who achieved neoadjuvant chemotherapy
* Confirmed operability with imaging study after neoadjuvant chemotherapy
* Age over 20 years old
* ECOG Performance status : 0-2
* The patient with written informed consent form

Exclusion Criteria:

* The patient with previous ipsilateral breast cancer history
* The patinet with previous ipsilateral axillary surgical procedure (e.g. excisional or incisional biopsy, axillary dissection)
* The patient without neoadjuvant chemotherapy
* Inoperable imaging study after neoadjuvant chemotherapy
* Inflammatory breast cancer
* Pregnant patient

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Identification rate of sentinel lymph node | during operation
  Collection of data for detection rate of sentinel lymph node for each group following direct comparison between each arms.

SECONDARY OUTCOMES:
Comparison of operation time for sentinel lymph node biopsy | during operation
  collection of data for operation time between skin incision and detection of sentinel lymph node, following direct comparison between each arms

CONTACTS AND LOCATIONS:
Overall Officials: Seeyoun Lee, Doctor, Principal Investigator — National Cancer Center, Korea
Locations (2):
- South Korea (2):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - National cancer center, Goyang-si, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data was generated on June 30, 2026, and can be provided for three years thereafter.
Access Criteria: a publication of a paper about this study